CLINICAL TRIAL: NCT06332573
Title: Impact of Onco-sexology Support on the Quality of Life of Patients Newly Diagnosed for Cancer
Acronym: SEXOCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-06
Record Dates: First submitted 2023-01-03; First posted 2024-03-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Early intervention" group (Experimental)
  Interventions: Other: Onco-sexology support
- "Late intervention" group (Other)
  Interventions: Other: Onco-sexology support

INTERVENTIONS:
Other: Onco-sexology support — Initiation of onco-sexology support before the introduction of systemic oncology treatment
  Arms: "Early intervention" group
Other: Onco-sexology support — Initiation of onco-sexology support after the introduction of systemic oncology treatment (2-3 months after the start of treatment).
  Arms: "Late intervention" group

SUMMARY:
Onco-sexology as a supportive care for patients treated for cancer is still rarely discussed or even non-existent in 2022. However, it's recommended to integrate the preservation of sexual health throughout the treatment and post-cancer process, given the impact of cancer, treatments and the importance of intimate life for a majority of patients.

Onco-sexology is one of the supportive care services validated by The French National Cancer Institute (INCa). It is also an objective of the 2014-2019 cancer plan and the 2017-2030 national sexual health strategy plan.

Although sexuality is one of the fundamental needs of the human being, including in the case of a chronic disease or cancer diagnosis, the lack of training of health professionals to deal with intimate life, the difficulty to exchange on this subject between caregivers and patients, the lack of financial support for onco-sexology consultations, are all obstacles to the global management of oncology patients. However, it's a request from patients to be able to discuss the subject in an intimate way with a professional.

While onco-sexology is already recommended as supportive care, a study on the impact of the delay in the management of sexual difficulties on quality of life could provide a sufficient level of evidence to change the practices and the care pathway of the oncology patient. Our objective is to study whether early management in onco-sexology has an impact on quality of life compared to late management (ie onco-sexology consultation before vs. after introduction of systemic oncological treatment).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Newly cancer diagnosis, including palliative care
* Having given free and informed written consent

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Persons deprived of their liberty by a judicial or administrative decision.
* Persons who are subject to a legal protection measure or who are unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-08-22 (Estimated); Study Completion 2028-01-22 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with improved quality of life as measured by the 36-Item Short Form Survey (SF-36) at the end of onco-sexology support | 4 months

SECONDARY OUTCOMES:
Evaluation of the quality of life of patients at 6 and 12 months after the end of onco-sexology support through the 36-Item Short Form Survey (SF-36) questionnaire | 6 and 12 months after the end of onco-sexology support
Evaluation of the quality of sexual life at the end of the onco-sexology support in both groups through specific questionnaires (The sexual quality of life-female and men) | 4 months
Evaluation of the quality of sexual life at 6 and 12 months after the end of the onco-sexology support through specific questionnaires (The sexual quality of life-female and men) | 6 and 12 months after the end of onco-sexology support
Evaluation of the body image, at the end of the onco-sexology support through the "Body Image Scale ". | 4 months
Evaluation of the body image, of the patient at 6 and 12 months after the last consultation with the onco-sexologist through the "Body Image Scale". | 6 and 12 months after the last consultation with the onco-sexologist
Evaluation of the satisfaction of the patient at the end of the care in onco-sexology care | 6 and 12 months after the end of onco-sexology support
Rate of patients expressing sexual difficulties during the consultation of announcement | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Européen Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No